CLINICAL TRIAL: NCT00519714
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Multi-Center Study to Evaluate the Lipid Regulating Effects of 1-Methylnicotinamide (1-MNA)
Brief Title: A Study to Evaluate the Lipid Regulating Effects of 1-Methylnicotinamide (1-MNA)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Commonwealth Medical Clinic (Unknown); Institut de Recherches Cliniques de Montreal (Other); Clinique des maladies lipidiques de Québec (Unknown); Centre de médecine genique communautaire (Unknown); Omnispec clinical research Inc (Unknown); Manna Research (Unknown); St. Jerome Medical Research Inc. (Other); Royal Victoria Hospital, Canada (Other); Hotel Dieu Hospital (Other); St Michael's Hospital Health Center (Unknown); Cambridge Cardiac Care Centre (Other); Maritime Research Center (Other); Rhodin Recherche Clinique (Unknown); Queen Elizabeth II Health Sciences Centre (Other); First Line Medical Ltd (Unknown); Diabetes Research, Vancouver General Hosp (Unknown); The Allin Clinic (Other); St Paul's Hospital Healthy Heart Clinical Trial (Unknown); The Clinical Trials Centre (Unknown); Recherche Invascor Inc (Other); MSHJ Research Associates (Other); Dr.Kim W Tan (Unknown)
Responsible Party: Jean-Claude Tardif/Researcher, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNAI-MNA-001
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — N(1)-methylnicotinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): three placebo capsules PO three times daily.
  Interventions: Dietary Supplement: Placebo
- 2 (Active Comparator): 1-MNA 90 mg daily: one active treatment capsule and two placebo capsules PO three times daily
  Interventions: Dietary Supplement: 1-Methylnicotinamide (1-MNA)
- 3 (Active Comparator): 1-MNA 270 mg daily: three active treatment capsules PO three times daily.
  Interventions: Dietary Supplement: 1-Methylnicotinamide (1-MNA)

INTERVENTIONS:
Dietary Supplement: 1-Methylnicotinamide (1-MNA) — Following a 6-8-week placebo and dietary-controlled baseline period, 195 men and women will be randomized to receive placebo, 30 mg MNA or 90 mg MNA three times daily for twelve weeks.
  Other Names: 1-MNA
  Arms: 2; 3
Dietary Supplement: Placebo — Placebo
  Arms: 1

SUMMARY:
A randomized, double-blind, placebo-controlled, dose-ranging, multi-center study. Following a 6-8 week placebo and dietary-controlled baseline period, approximately 195 men and women with either hypertriglyceridemia or mixed hyperlipidemia with serum triglycerides (TG) > 200 mg/dl (2.26 mmol/l) will be randomized to receive either placebo, 30 mg 1-MNA or 90 mg 1-MNA three times daily for twelve weeks. Lipid and ancillary exploratory parameters will be evaluated at screening, during the baseline period, upon randomisation and throughout the 12-week active treatment period. Additionally, blood samples will be drawn at randomisation and at clinic visits during the active treatment period for sparse sampling population pharmacokinetic assessments. All blood samples for lipid assessments and glucose measurements will be collected following a 12-hour fast. Safety and tolerability will be assessed throughout the trial through the evaluation of physical exams, ECGs, routine hematology and blood chemistry testing, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age at the time of informed consent (women of childbearing potential must be practicing adequate contraception)
* Patients with mean serum TG > 200 mg/dl (2.26 mmol/l) and < 700 mg/dl (7.91 mmol/l) as measured at 2 sequential visits during the dietary controlled baseline period (Visits 2 and 3 or Visits 3 and 3a) and having lower level within 25% of upper level (higher value minus lower value)/higher value < 0.25)
* Patients willing and able to sign an informed consent form and follow the protocol

Exclusion Criteria:

* Patients who are pregnant or nursing
* Patients with evidence of hepatic (ALT or AST greater than 1.5 ULN, bilirubin greater than 1.5 ULN, or cirrhosis) or renal dysfunction (serum creatinine greater than 140 μmol/l, or nephrotic syndrome) as measured during the baseline phase
* Patients with uncontrolled diabetes mellitus (fasting glucose level above 11 mmol/l or HbA1C above 10%) as measured during the baseline phase
* Patients with hypothyroidism that is not treated or not stable for at least 6 months prior to study entry
* Patients with uncontrolled hypertension (systolic blood pressure above 160 mm Hg and/or diastolic blood pressure above 110 mm Hg)
* Patients with systolic blood pressure above 140 mm Hg AND three or more of the following cardiovascular risk factors:

  * Current cigarette smoker
  * HDL-C < 40 mg/dL (1.04 mmol/L)
  * Coronary heart disease in male first degree relative < 55 years of age
  * Coronary heart disease in female first degree relative < 65 years of age
  * Male age 45 years or older
  * Female age 55 years or older
* Patients with known hyperuricemia or with a history of gout
* Patients with an active peptic ulcer
* Patients with known coronary artery disease, cerebrovascular disease or peripheral arterial disease that has previously required PCI or surgical intervention
* Patients with known intolerance or allergy to niacin
* Patients consuming more than 10 alcoholic drinks per week
* Patients with a history of drug abuse
* Patients receiving any lipid modifying agent within 4 weeks of entry into the baseline period
* Patients participating in another clinical trial within 30 days of entry into the baseline period
* Patients considered to be non-compliant to study medication (< 80% study medication) or diet during the placebo-baseline phase
* Patients for whom the investigator determines that the study would not be appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The percent change in total serum Triglycerides from baseline to end of study | 12 weeks

SECONDARY OUTCOMES:
The percent change in total cholesterol, low-density lipoprotein cholesterol, very low-density lipoprotein cholesterol, high-density lipoprotein cholesterol , total apolipoprotein B , apolipoprotein A1 and TG/HDL-C ratio from baseline to end of study. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Institut de Cardiologie de Montreal, Montreal, Quebec, Canada